CLINICAL TRIAL: NCT01075256
Title: An Exploratory Clinical Study to Evaluate the Efficacy of Two Currently Marketed Toothpastes Containing Different Concentrations of a Tubule Occlusion Agent
Brief Title: Dose Response of a Tubule Occlusion Agent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z3690607
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-04

CONDITIONS: Dentine Hypersensitivity; Dental Pain
Keywords: sensitivity; occlusion
MeSH Terms: conditions — Dentin Sensitivity; Toothache; Hypersensitivity; Bites and Stings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5% calcium sodium phosphosilicate toothpaste (Active Comparator): Participants to brush their teeth for two minutes, twice daily for 15 days with 5% sodium calcium phosphosilicate toothpaste.
  Interventions: Device: 5% calcium sodium phosphosilicate toothpaste
- 7.5% calcium sodium phosphosilicate toothpaste (Active Comparator): Participants to brush their teeth for two minutes, twice daily for 15 days with 7.5% sodium calcium phosphosilicate toothpaste.
  Interventions: Device: 7.5% calcium sodium phosphosilicate toothpaste
- Placebo toothpaste (Placebo Comparator): Participants to brush their teeth for two minutes, twice daily for 15 days with placebo toothpaste.
  Interventions: Device: Placebo toothpaste

INTERVENTIONS:
Device: 5% calcium sodium phosphosilicate toothpaste — Low concentration calcium sodium phosphosilicate tubule occlusion agent
  Arms: 5% calcium sodium phosphosilicate toothpaste
Device: 7.5% calcium sodium phosphosilicate toothpaste — High concentration calcium sodium phosphosilicate tubule occlusion agent
  Arms: 7.5% calcium sodium phosphosilicate toothpaste
Device: Placebo toothpaste — Placebo toothpaste
  Arms: Placebo toothpaste

SUMMARY:
To evaluate the efficacy of two different concentrations of a tubule occlusion agent - calcium sodium phosphosilicate in treatment of dentine hypersensitivity

DETAILED DESCRIPTION:
Dentine hypersensitivity is characterized by short, sharp pain arising from exposed dentine typically in response to chemical, thermal, tactile or osmotic stimuli. Dentine hypersensitivity may be treated by either making the nerve in the tooth less sensitive or by occluding the tubules to limit exposure of the nerve to external stimuli. Bioactive and biocompatible glasses react with oral fluid to deposit a mineral that is chemically analogous to that found in both enamel and dentine thus preventing exposure of the nerve to external stimuli.

A number of controlled clinical trials have been reported indicating that a calcium sodium phosphosilicate bioactive glass, when incorporated into a toothpaste formulation, significantly reduce pain from dentine hypersensitivity. The aim of this study is to evaluate the effectiveness of two currently marketed toothpastes, containing 5% calcium sodium phosphosilicate and the other containing 7.5% calcium sodium phosphosilicate in the treatment of dentine hypersensitivity compared to a matched placebo control.

ELIGIBILITY:
Inclusion Criteria:

1. Consent: Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
2. Age: Aged between 20 - 50 years.
3. General Health: Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history.
4. Contraception: Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception.
5. Erosion/Abrasion/Recession:Study teeth must show signs of facial/cervical erosion, abrasion and/or gingival recession.
6. Gingival Health / Tooth Mobility Grade:Study teeth must have Löe and Silness Gingival Index (GI) score less than or equal to 2 and clinical mobility less than or equal to grade I.
7. Current Product Use: Participants must have been using the same brand of toothpaste for at least 2 months and should not have used desensitizing toothpaste during the 4 weeks preceding screening. Participants will be required to bring in their current toothpaste(s) in order to verify the ingredients.
8. VAS Training: Successfully completes the VAS training exercise at Screening.
9. Sensitivity: Self-reported history of dentinal hypersensitivity and a primary complaint of sensitive teeth lasting a maximum of 10 years. At Screening: A minimum of 5 evaporative (air) sensitive lateral incisors, canines or pre-molars must display a response greater than 25 mm on a 100 mm VAS. At Baseline: A minimum of 3 of the 5 evaporative (air) sensitive teeth identified at screening must display a response greater than 25 mm on a 100 mm VAS. All teeth meeting the sensitivity Inclusion Criteria will be followed and assessed using both efficacy parameters.
10. Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions.

Exclusion Criteria:

1. Pregnancy: Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
2. Breast-feeding: Women who are breast-feeding.
3. Medical History: a) Chronic debilitating disease is present b)Chronic disease or other condition is present that is associated with intermittent episodes or constant daily pain, such as arthritis, low back pain, dysmenorrhea, etc.
4. Medications: Daily doses of medication, which in the opinion of the investigator, might interfere with the perception of pain, are being taken. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, mood-altering and anti-inflammatory drugs.
5. Dentition Exclusions: a) Sensitive teeth not expected to respond to treatment with an over-the- counter (OTC) dentifrice in the opinion of the investigator. b) Teeth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns, orthodontic bands, extensive caries or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine. c) Dental professional hygiene (includes dental prophylaxis, irrigation, and intensive anti-microbial/anti-biotic therapy) within 14 days of the screening visit. d) Presence of dental implants. e) Lip or tongue piercings. f) Periodontal surgical history within the past 6 months or have been scaled /root planed within the past 3 months.
6. Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
7. Clinical Study/Experimental Medication: a) Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.b) Previous participation in this study.
8. Xerostomia: Any condition or medication that causes xerostomia.
9. Personnel: An employee of the sponsor or the study site or members of their immediate family.
10. Other: Any subject who in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- University Park Research Center (UPRC), Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: During the first 4 weeks of the study all participants brushed with an acclimatization toothpaste (sodium fluoride [NaF] toothpaste containing 1100 parts per million [ppm] fluoride [F]) for maintaining wash-out period and standardizing the oral conditions.
Groups:
- 7.5% Sodium Calcium Phosphosilicate Toothpaste: Participants brushed their teeth for two minutes, twice daily for 15 days with 7.5% sodium calcium phosphosilicate toothpaste. All study treatments were fluoride free.
- 5% Sodium Calcium Phosphosilicate Toothpaste: Participants brushed their teeth for two minutes, twice daily for 15 days with 5% sodium calcium phosphosilicate toothpaste. All study treatments were fluoride free.
- Placebo Toothpaste: Participants brushed their teeth for two minutes, twice daily for 15 days with a sodium calcium phosphosilicate free placebo toothpaste. All study treatments were fluoride free.
Period: Overall Study
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Started | 64 | 66 | 65
Completed | 63 | 66 | 65
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Sodium Calcium Phosphosilicate Toothpaste | 7.5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste | Total
Number analyzed (Participants) | 66 | 63 | 66 | 195
Age Continuous [Mean (Standard Deviation); unit: years] | 38.30 (8.925) | 37.63 (8.920) | 36.61 (9.885) | 37.51 (9.239)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population reported as treated- one randomized participant in the High concentration group received placebo and is included in the placebo count.
  Participants
    Female | 51 | 49 | 54 | 154
    Male | 15 | 14 | 12 | 41

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Evaporative Air Sensitivity Pain Response on a Visual Analog Scale (VAS) at Day 15
Description: Response to a constant jet of air applied to a hypersensitive tooth was evaluated using a 100 millimeter (mm) VAS pain response scale. According to this analog scale, pain response for stimulated tooth ranged from 0 (no pain) to 100 (intense pain). Change from baseline in pain response was calculated using VAS score and a change of greater than 25 mm in VAS indicates potential relevant clinical significance of treatment.
Time Frame: Baseline to Day 15
Population: Intention to treat (ITT) population: All randomized participants who received at least one dose of investigational product who have at least one post-baseline efficacy measure. Missing data was not imputed. Due to drop outs, there was difference in number of participants analyzed.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 63 | 66 | 65
Units on a scale | -26.1 [-29.40 to -22.72] | -28.4 [-31.60 to -25.12] | -26.2 [-29.54 to -22.95]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; The null hypothesis was no diference between treatments in comparison. Statistical tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.3628, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -2.1, 95% CI 2-sided [-6.70 to 2.46] — Difference was first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; The null hypothesis was no difference between treatments in comparison. Statistical tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.9361, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 0.2, 95% CI 2-sided [-4.45 to 4.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3257, ANCOVA — No adustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean difference = 2.3, 95% CI 2-sided [-2.31 to 6.92] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment

2. Secondary Outcome: Adjusted Mean Change From Baseline in Evaporative Air Sensitivity Pain Response on a VAS at Day 7
Description: as for outcome 1
Time Frame: Baseline to Day 7
Population: ITT population: All randomized participants who received at least one dose of investigational product who have at least one post-baseline efficacy measure. Missing data was not imputed. Due to drop outs, there was difference in number of participants analyzed.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- 7.5% Sodium Calcium Phosphosilicate Toothpaste: Participants brushed their teeth for two minutes, twice daily with 7.5% sodium calcium phosphosilicate toothpaste. All study treatments were fluoride free.
- 5% Sodium Calcium Phosphosilicate Toothpaste: Participants brushed their teeth for two minutes, twice daily with 5% sodium calcium phosphosilicate toothpaste. All study treatments were fluoride free.
- Placebo Toothpaste: Participants brushed their teeth for two minutes, twice daily with a sodium calcium phosphosilicate free placebo toothpaste. All study treatments were fluoride free.
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 63 | 66 | 65
Units on a scale | -16.4 [-19.80 to -12.93] | -17.4 [-20.75 to -14.10] | -16.4 [-19.78 to -13.02]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6674, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -1.0, 95% CI 2-sided [-5.73 to 3.68] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9888, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 0.0, 95% CI 2-sided [-4.74 to 4.81] — Difference is the high concentration minus placebo such that a positive difference favors the first named treatment
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6599, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 1.1, 95% CI 2-sided [-3.69 to 5.81] — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Adjusted Mean Change From Baseline in Cold Water Sensitivity Pain Response on a VAS at Day 15
Description: Response of exposed dentine surface to application of 1 ml freshly melted ice cold water was evaluated using a 100 mm VAS pain response scale. According to this analog scale, pain response for stimulated tooth ranged from 0 (no pain) to 100 (intense pain). Change from baseline in pain response was calculated using VAS score and a change of greater than 25 mm in VAS indicates potential relevant clinical significance of treatment.
Time Frame: Baseline to Day 15
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 63 | 66 | 65
Units on a scale | -32.8 [-37.55 to -28.00] | -32.2 [-36.86 to -27.59] | -32.3 [-37.04 to -27.60]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9759, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 0.1, 95% CI 2-sided [-6.34 to 6.54] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8903, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -0.5, 95% CI 2-sided [-6.97 to 6.06] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment; Test type: Superiority or Other; p = 0.8662, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted mean difference = -0.6, 95% CI 2-sided [-7.04 to 5.93] — [estimate comment as in outcome 1, analysis 3]

4. Secondary Outcome: Adjusted Mean Change From Baseline in Cold Water Sensitivity Pain Response on a VAS at Day 7
Description: as for outcome 3
Time Frame: Baseline to Day 7
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 63 | 66 | 65
Units on a scale | -21.5 [-26.14 to -16.81] | -22.5 [-26.99 to -17.93] | -21.8 [-26.44 to -17.21]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; Null hypothesis was no difference between treatments in comparison. Statistical tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.8419, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -0.6, 95% CI 2-sided [-6.93 to 5.66] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9147, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 0.3, 95% CI 2-sided [-6.03 to 6.72] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7600, ANCOVA — No adjustments for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 1.0, 95% CI 2-sided [-5.36 to 7.33] — [estimate comment as in outcome 1, analysis 3]

5. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in Evaporative Air Sensitivity Pain Response on a VAS at Day 10
Description: Response to a constant jet of air applied to a hypersensitive tooth was evaluated using a 100mm VAS pain response scale. According to this analog scale, pain response for stimulated tooth ranged from 0 (no pain) to 100 (intense pain). Change from baseline in pain response was calculated using VAS score and a change of greater than 25 mm in VAS indicates potential relevant clinical significance of treatment.
Time Frame: Baseline to Day 10
Population: ITT population subset: A subset of randomized participants who received at least one dose of investigational product who have at least one post-baseline efficacy measure. Missing data was not imputed. Due to drop outs, there was difference in number of participants analyzed.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Placebo Toothpaste: Participants brushed their teeth for two minutes, twice daily with a sodium calcium phosphosilicate (NovaMin) free placebo toothpaste. All study treatments were fluoride free.
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 18 | 18 | 17
Units on a scale | -28.7 [-34.90 to -22.43] | -22.7 [-33.70 to -21.67] | -28.2 [-34.46 to -21.88]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9124, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 0.5, 95% CI 2-sided [-8.28 to 9.24] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9083, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -0.5, 95% CI 2-sided [-9.13 to 8.14] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.8231, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -1.0, 95% CI 2-sided [-9.73 to 7.77] — [estimate comment as in outcome 1, analysis 3]

6. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in Cold Water Sensitivity Pain Response on a VAS at Day 10
Description: as for outcome 3
Time Frame: Baseline to Day 10
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Placebo Toothpaste: Participants brushed their teeth for two minutes, twice daily with sodium calcium phosphosilicate free placebo toothpaste. All study treatments were fluoride free.
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 18 | 18 | 17
Units on a scale | -34.7 [-44.24 to -25.09] | -31.3 [-40.03 to -22.62] | -34.7 [-44.22 to -25.21]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5946, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 3.4, 95% CI 2-sided [-9.32 to 16.09] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9944, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 0.0, 95% CI 2-sided [-12.51 to 12.60] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5998, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -3.3, 95% CI 2-sided [-16.06 to 9.38] — [estimate comment as in outcome 1, analysis 3]

7. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in Evaporative Air Sensitivity Pain Response on a VAS at Day 3
Description: Response to a constant jet of air applied to a hypersensitive tooth was evaluated using a 100 mm VAS pain response scale. According to this analog scale, pain response for stimulated tooth ranged from 0 (no pain) to 100 (intense pain). Change from baseline in pain response was calculated using VAS score and a change of greater than 25 mm in VAS indicates potential relevant clinical significance of treatment.
Time Frame: Baseline to Day 3
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 18 | 18 | 17
Units on a scale | -13.5 [-20.08 to -6.87] | -12.3 [-18.66 to -5.90] | -11.1 [-17.74 to -4.40]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7952, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-10.51 to 8.09] — Difference is first named treatment minus second named treatment such that a positive difference favours the first named treatment
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6010, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -2.4, 95% CI 2-sided [-11.56 to 6.76] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7976, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-10.48 to 8.10] — [estimate comment as in outcome 1, analysis 3]

8. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in Cold Water Sensitivity Pain Response on a VAS at Day 3
Description: as for outcome 3
Time Frame: Baseline to Day 3
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Number analyzed (Participants) | 18 | 18 | 17
Units on a scale | -19.3 [-27.56 to -11.02] | -16.9 [-24.44 to -9.44] | -17.6 [-25.79 to -9.40]
Statistical Analysis 1: Comparison: 5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9060, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = 0.7, 95% CI 2-sided [-10.38 to 11.68] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs Placebo Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7575, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -1.7, 95% CI 2-sided [-12.63 to 9.25] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: 7.5% Sodium Calcium Phosphosilicate Toothpaste vs 5% Sodium Calcium Phosphosilicate Toothpaste; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6727, ANCOVA — No adjustment was made for multiple comparisons; ANCOVA model adjusted for baseline, treatment and number of sensitive teeth and years of sensitivity; Adjusted Mean Difference = -2.3, 95% CI 2-sided [-13.42 to 8.73] — [estimate comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | 7.5% Sodium Calcium Phosphosilicate Toothpaste | 5% Sodium Calcium Phosphosilicate Toothpaste | Placebo Toothpaste
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 3/63 | 3/66 | 3/66
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7.5% Sodium Calcium Phosphosilicate Toothpaste (N=63) | 5% Sodium Calcium Phosphosilicate Toothpaste (N=66) | Placebo Toothpaste (N=66)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Gingival Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Mouth Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinus Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
An issue with study product packaging was discovered post-study completion. The nature indicated that subject response was likely to have been liable to a positive bias. Efficacy cannot be considered as valid and no reliable conclusions possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No